CLINICAL TRIAL: NCT05182307
Title: Use of DurAVR™ THV System in Subjects With Severe Aortic Stenosis: First In Human Study
Brief Title: DurAVR™ THV System: First-In-Human Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anteris Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SP0011
Record Dates: First submitted 2021-12-06; First posted 2022-01-10 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Symptomatic Aortic Stenosis; Severe Aortic Valve Stenosis; Aortic Valve Calcification
Keywords: TAVI; TAVR; Transcatheter Aortic Valve Implantation; Transcatheter valve
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve, Calcification of

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): DurAVR™ THV System
  Interventions: Device: DurAVR™ THV System

INTERVENTIONS:
Device: DurAVR™ THV System — Transcatheter Aortic Valve Implantation (TAVI) Procedure

SUMMARY:
A prospective, non-randomized, single-arm, single-center, first-in-human study designed to evaluate the safety and feasibility of the DurAVR™ THV System in the treatment of subjects with symptomatic severe aortic stenosis.

DETAILED DESCRIPTION:
The DurAVR™ THV System is a novel balloon-expandable single-piece 3D transcatheter aortic valve.

The study will enroll up to 25 subjects suffering from severe, symptomatic aortic stenosis as determined by a Heart Team. Subjects will be consented for follow-up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic, severe aortic stenosis
2. Eligible for delivery of the DurAVR™ THV
3. Anatomy appropriate to accommodate safe placement of DurAVR™ THV
4. Understands the study requirements and the treatment procedures and provides written informed consent.
5. Subject agrees to complete all required scheduled follow-up visits.

Exclusion Criteria:

Anatomical

1. Anatomy precluding safe placement of DurAVR™ THV
2. Pre-existing prosthetic heart valve in any position
3. Unicuspid or bicuspid aortic valve
4. Severe aortic regurgitation
5. Severe mitral or severe tricuspid regurgitation requiring intervention
6. Moderate to severe mitral stenosis
7. Hypertrophic obstructive cardiomyopathy
8. Echocardiographic evidence of intracardiac mass, thrombus or vegetation requiring treatment
9. Severe basal septal hypertrophy with outflow gradient Clinical
10. Evidence of an acute myocardial infarction ≤ 30 days before the intended treatment
11. Determined inoperable/ineligible for surgery by the Heart Team
12. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to the index procedure
13. Blood dyscrasias as defined: leukopenia (WBC < 1000mm3), thrombocytopenia (platelet count < 50,000 cells/mm3), history of bleeding diathesis or coagulopathy, or hypercoagulable states
14. Untreated clinically significant Coronary Artery Disease (CAD) requiring revascularization
15. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support
16. Need for emergency surgery for any reason
17. Ventricular dysfunction with left ventricular ejection fraction (LVEF) ≤ 40% as measured by resting echocardiogram
18. Recent (within 6 months) cerebrovascular accident (CVA) or transient ischemic attack (TIA)
19. Symptomatic carotid or vertebral artery disease
20. End stage renal disease requiring chronic dialysis or creatinine clearance < 20 cc/min
21. GI bleeding within the past 3 months
22. A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated: aspirin, heparin, nitinol (titanium or nickel), ticlopidine and clopidogrel, contrast media
23. Ongoing sepsis, including active endocarditis
24. Subject refuses a blood transfusion
25. Life expectancy < 12 months due to associated non-cardiac co-morbid conditions
26. Other medical, social, or psychological conditions that in the opinion of an Investigator precludes the subject from appropriate consent
27. Severe dementia (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits)
28. Currently participating in an investigational drug or another investigational device trial
29. Subject belongs to a vulnerable population.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
DurAVR™ prosthetic heart valve implant | Immediate post procedure
  Number of subjects for which a single DurAVR™ prosthetic heart valve was correctly positioned into the proper anatomical location
Hemodynamic performance | Immediate post procedure
  Effective Orifice Area (EOA), Mean gradient, Aortic Regurgitation, Paravalvular Leak (PVL), Doppler Velocity Index (DVI)
All-cause mortality | 30 days
  All-cause mortality
All-cause mortality | 1 year
  All-cause mortality
Myocardial infarction | 30 days
  Myocardial infarction
Myocardial infarction | 1 year
  Myocardial infarction
Stroke | 30 days
  Disabling Stroke (VARC-3 Guidelines)
Stroke | 1 year
  Disabling Stroke (VARC-3 Guidelines)
Life-threatening bleeding | 30 days
  Life-threatening bleeding (VARC-3 Guidelines)
Life-threatening bleeding | 1 year
  Life-threatening bleeding (VARC-3 Guidelines)

OTHER OUTCOMES:
DurAVR™ THV System ease of use | Intra-operative
  DurAVR™ THV System ease of use (Questionnaire)
Adverse Events | Throughout the entire study, up to 1 year.
  VARC-3 defined adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Chris Meduri, MD, Study Director — Anteris Technologies
Locations (1):
- Tbilisi Heart and Vascular Clinic Ltd, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No